CLINICAL TRIAL: NCT04245202
Title: Comparison of High Flow Nasal Cannula and Standard Face Mask Oxygen Therapy in Children With Moderate and Severe Bronchiolitis; a Randomized Controlled Trial
Brief Title: Comparison of High Flow Nasal Cannula and Standard Face Mask Oxygen Therapy in Children With Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Aykut Eşki, Medical Doctor, Pediatric Pulmonology, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-TIP-012
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Acute Bronchiolitis
Keywords: Acute Bronchiolitis; High Flow Nasal Cannula; Standard Face Mask

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: HFNCOT (Active Comparator): Set between 2 to 25 l/min, adjusted to obtain peripheral oxygen saturation >92%.
  Interventions: Device: HFNCOT
- Active Comparator: St-FMOT (Active Comparator): To obtain oxygen saturation >92%
  Interventions: Other: St-FMOT

INTERVENTIONS:
Device: HFNCOT — The patient will receive a high flow nasal of humidified oxygen, set between 2 to 25 l/min. The inspired fraction of oxygen (FiO2) will be adjusted to obtain the oxygen saturation >92%.
  Arms: Active Comparator: HFNCOT
Other: St-FMOT — The inspired fraction of oxygen (FiO2) will be adjusted to obtain the oxygen saturation >92%.
  Arms: Active Comparator: St-FMOT

SUMMARY:
The study aims to compare the efficacy of two different oxygenation methods on decrease respiratory rate, heart rate, and clinical respiratory score in children with moderate to severe bronchiolitis requiring oxygen therapy.

1. Standard face mask oxygen therapy (St-FMOT)
2. High-flow nasal cannula oxygen therapy (HFNCOT)

DETAILED DESCRIPTION:
Bronchiolitis is the most common cause of hospitalization for children under one year of age and, caused by respiratory viruses. Although several medications and interventions studied for bronchiolitis treatment, hydration and oxygenation are the main treatments. High-flow nasal cannula oxygen therapy (HFNCOT) has been widely used to provide respiratory support in children with acute respiratory diseases.

Patients had earlier improvement with HFNCOT to decrease the respiratory rate and respiratory effort than patients with standard low-flow oxygen therapy (SOT).

HFNCOT therapy reduced more effective in heart rate, respiratory effort, and length of supportive oxygen treatment (LOOT) compared with SOT. However, the length of hospital stay (LOS) and feeding ability had better consequences in patients with moderate and severe bronchiolitis treated with HFNCOT.

Another published study shows that in infants with acute bronchiolitis, which required oxygen therapy, there was no significant difference between therapy groups in terms of LOOT, LOS, and admission to the intensive care unit (ICU). HFNCOT was more efficient than SOT and reduced the rate of intubation/invasive ventilation in severe bronchiolitis management. Despite these beneficial effects of HFNCOT, it was not recommended by international guidelines yet. However, well designed, prospective randomized controlled trials are still needed to use this therapy in the wards.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1-24 months applied with moderate and severe bronchiolitis requiring supplemental oxygen were eligible for the study.
* The severity of bronchiolitis was assessed according to the clinical respiratory score (CRS) of Liu et al. (5). The patients with CRS ≥5 were included.
* Peripheral oxyhemoglobin saturation is < 92%.

Exclusion criteria:

* Children admitted to the ICU for urgent invasive mechanical ventilation;
* those who received standard oxygen therapy (SOT) or HFNCOT at other facilities before arrival;
* those with an underlying medical condition (such as congenital heart disease, chronic lung disease, neuromuscular disease, metabolic disease, or immunocompromised);
* those who had a craniofacial malformation, an upper airway obstruction, pneumothorax, or nasal trauma, and missing parental consent or a refused permission of the participant.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aykut Eşki, MD, Principal Investigator — Ege University Medical Study
Locations (1):
- Ege University Medical Faculty, Izmir, Select A State, Turkey (Türkiye)

REFERENCES:
- [Result] Franklin D, Babl FE, Schlapbach LJ, Oakley E, Craig S, Neutze J, Furyk J, Fraser JF, Jones M, Whitty JA, Dalziel SR, Schibler A. A Randomized Trial of High-Flow Oxygen Therapy in Infants with Bronchiolitis. N Engl J Med. 2018 Mar 22;378(12):1121-1131. doi: 10.1056/NEJMoa1714855. PMID 29562151
- [Result] Franklin D, Dalziel S, Schlapbach LJ, Babl FE, Oakley E, Craig SS, Furyk JS, Neutze J, Sinn K, Whitty JA, Gibbons K, Fraser J, Schibler A; PARIS and PREDICT. Early high flow nasal cannula therapy in bronchiolitis, a prospective randomised control trial (protocol): A Paediatric Acute Respiratory Intervention Study (PARIS). BMC Pediatr. 2015 Nov 14;15:183. doi: 10.1186/s12887-015-0501-x. PMID 26572729
- [Result] Liu G, Fan C, Wu H. High-flow nasal cannula therapies for respiratory management in pediatric patients. Minerva Pediatr. 2018 Oct;70(5):488-492. doi: 10.23736/S0026-4946.17.04781-8. Epub 2017 Mar 27. PMID 28353318
- [Result] Pham TM, O'Malley L, Mayfield S, Martin S, Schibler A. The effect of high flow nasal cannula therapy on the work of breathing in infants with bronchiolitis. Pediatr Pulmonol. 2015 Jul;50(7):713-20. doi: 10.1002/ppul.23060. Epub 2014 May 21. PMID 24846750
- [Result] Bressan S, Balzani M, Krauss B, Pettenazzo A, Zanconato S, Baraldi E. High-flow nasal cannula oxygen for bronchiolitis in a pediatric ward: a pilot study. Eur J Pediatr. 2013 Dec;172(12):1649-56. doi: 10.1007/s00431-013-2094-4. Epub 2013 Jul 31. PMID 23900520
- [Result] Milesi C, Pierre AF, Deho A, Pouyau R, Liet JM, Guillot C, Guilbert AS, Rambaud J, Millet A, Afanetti M, Guichoux J, Genuini M, Mansir T, Bergounioux J, Michel F, Marcoux MO, Baleine J, Durand S, Durand P, Dauger S, Javouhey E, Leteurtre S, Brissaud O, Renolleau S, Portefaix A, Douillard A, Cambonie G; GFRUP Respiratory Study Group. A multicenter randomized controlled trial of a 3-L/kg/min versus 2-L/kg/min high-flow nasal cannula flow rate in young infants with severe viral bronchiolitis (TRAMONTANE 2). Intensive Care Med. 2018 Nov;44(11):1870-1878. doi: 10.1007/s00134-018-5343-1. Epub 2018 Oct 21. PMID 30343318
- [Result] Mace AO, Gibbons J, Schultz A, Knight G, Martin AC. Humidified high-flow nasal cannula oxygen for bronchiolitis: should we go with the flow? Arch Dis Child. 2018 Mar;103(3):303. doi: 10.1136/archdischild-2017-313950. Epub 2017 Sep 13. No abstract available. PMID 28903952
- [Result] Testa G, Iodice F, Ricci Z, Vitale V, De Razza F, Haiberger R, Iacoella C, Conti G, Cogo P. Comparative evaluation of high-flow nasal cannula and conventional oxygen therapy in paediatric cardiac surgical patients: a randomized controlled trial. Interact Cardiovasc Thorac Surg. 2014 Sep;19(3):456-61. doi: 10.1093/icvts/ivu171. Epub 2014 Jun 8. PMID 24912486
- [Result] Milesi C, Boubal M, Jacquot A, Baleine J, Durand S, Odena MP, Cambonie G. High-flow nasal cannula: recommendations for daily practice in pediatrics. Ann Intensive Care. 2014 Sep 30;4:29. doi: 10.1186/s13613-014-0029-5. eCollection 2014. PMID 25593745
- [Result] Schibler A, Franklin D. Respiratory support for children in the emergency department. J Paediatr Child Health. 2016 Feb;52(2):192-6. doi: 10.1111/jpc.13078. PMID 27062623
- [Result] Da Dalt L, Bressan S, Martinolli F, Perilongo G, Baraldi E. Treatment of bronchiolitis: state of the art. Early Hum Dev. 2013 Jun;89 Suppl 1:S31-6. doi: 10.1016/S0378-3782(13)70011-2. PMID 23809346
- [Result] Beggs S, Wong ZH, Kaul S, Ogden KJ, Walters JA. High-flow nasal cannula therapy for infants with bronchiolitis. Cochrane Database Syst Rev. 2014 Jan 20;2014(1):CD009609. doi: 10.1002/14651858.CD009609.pub2. PMID 24442856
- [Derived] Eski A, Ozturk GK, Turan C, Ozgul S, Gulen F, Demir E. High-flow nasal cannula oxygen in children with bronchiolitis: A randomized controlled trial. Pediatr Pulmonol. 2022 Jun;57(6):1527-1534. doi: 10.1002/ppul.25893. Epub 2022 Mar 28. PMID 35293153

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From March 14, 2017, through March 10, 2020, 5643 patients were presented to the emergency department and pediatric pulmonology unit of Ege University Medical Faculty. Four hundred seventy-two children were eligible for the study, with 134 missing opportunities to enroll, and 251 parents declined consent. We randomly assigned 87 children to Standard face mask oxygen therapy and High-Flow nasal cannula therapy.
Pre-assignment Details: No patients were excluded from the study after participant enrollment.
Groups:
- St-FMOT: Children in the standard-therapy group received supplemental oxygen via a simple face mask, a range of 6-10 L/min, to maintain oxygen saturation level between 92-98%. Those who sustained the oxygen saturation >92% in the ambient oxygen concentration were weaned off Standard face mask oxygen therapy.
- HFNCOT: Children in the high-flow group received heated and humidified high-flow oxygen at a rate of 2 L*kg/min (maximum 25 L/min), using an age-appropriate Optiflow Junior cannula and Airvo 2 high-flow system (Fisher and Paykel Healthcare). The initial fraction of inspired oxygen (FiO2) was set at 40%. The starting flow rate continued for a minimum of 4 hours. According to the patients' clinical response, the flow rate was decreased by 0.5 L*kg/min per hour. The FiO2 was adjusted to obtain the oxygen saturation levels between 92-98%. When the flow rate was at 0.5 L*kg/min, and the FiO2 was equal to the ambient oxygen concentration, High-Flow nasal cannula oxygen therapy was stopped.
Period: Overall Study
Arm/Group | St-FMOT | HFNCOT
Started | 48 (After getting consent.) | 39 (After getting consent)
Completed | 38 | 38
Not Completed | 10 | 1
Not completed — Lack of Efficacy | 10 | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographic characteristics of participants according to allocation (Intention-to-treat analysis)
Groups:
- St-FMOT: Children who received standard face mask oxygen treatment
- HFNCOT: Children who received high flow nasal cannula oxygen treatment
- Total: Total of all reporting groups
Arm/Group | St-FMOT | HFNCOT | Total
Number analyzed (Participants) | 48 | 39 | 87
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 6.5 [3.6 to 11.0] | 6.0 [3.0 to 12.0] | 6.0 [3.5 to 11.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 27 | 24 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Turkey | 48 | 39 | 87
Gestational age at birth [Count of Participants; unit: Participants]
  Prematurity (< 37 weeks) | 7 | 8 | 15
  Term infant (> 36 weeks) | 41 | 31 | 72
Weight at the admission (kg) [Median (Inter-Quartile Range); unit: kilogram] | 7.4 [6.0 to 9.5] | 8.0 [5.1 to 10.0] | 8.0 [6.0 to 9.7]
Baseline heart rate [Median (Inter-Quartile Range); unit: beat per minute] | 174.0 [156.2 to 186.5] | 170.0 [157.0 to 188.0] | 173.0 [157.0 to 188.0]
Baseline respiratory rate [Median (Inter-Quartile Range); unit: Breaths per minute] | 64.5 [60.0 to 70.0] | 66.0 [60.0 to 72.0] | 66.0 [60.0 to 70.0]
Baseline Oxygen Saturation [Median (Inter-Quartile Range); unit: percentage of saturated oxygen] | 88.0 [86.2 to 89.0] | 87.0 [84.0 to 88.0] | 88.0 [86.0 to 88.0]
Baseline clinical respiratory score [Median (Inter-Quartile Range); unit: score on a scale] — Unabbreviated scale title: Clinical Respiratory Score, categorizing as severe bronchiolitis (9-12 points), moderate bronchiolitis (5-8 points), and mild bronchiolitis (0-4 points). Higher scores mean a worse outcome. This score involves respiratory rate, retraction, dyspnea/consciousness status, and wheezing. Each variable ranges from 0 to 3 points.
  score on a scale | 9.0 [7.0 to 10.2] | 9.5 [8.7 to 11.0] | 9.0 [8.0 to 11.0]
Severity of clinical respiratory score [Count of Participants; unit: Participants] — Unabbreviated scale title: Clinical Respiratory Score, categorizing as severe bronchiolitis (9-12 points), moderate bronchiolitis (5-8 points), and mild bronchiolitis (0-4 points). Higher scores mean a worse outcome. This score involves respiratory rate, retraction, dyspnea/consciousness status, and wheezing. Each variable ranges from 0 to 3 points.
  Participants
    Moderate | 18 | 9 | 27
    Severe | 30 | 30 | 60
Season admitted [Count of Participants; unit: Participants]
  Winter | 28 | 25 | 53
  Autumn | 9 | 7 | 16
  Spring | 7 | 4 | 11
  Summer | 4 | 3 | 7
Number of detected virus [Count of Participants; unit: Participants]
  No virus | 2 | 0 | 2
  1 virus | 39 | 32 | 71
  2 viruses | 7 | 7 | 14
Virus detected [Count of Participants; unit: Participants]
  RSV | 19 | 21 | 40
  HRV | 7 | 4 | 11
  FLUA | 2 | 1 | 3
  PIV3 | 1 | 1 | 2
  HBoV | 4 | 3 | 7
  hMPV | 4 | 2 | 6
  hCoV | 0 | 0 | 0
  RSV+HRV | 0 | 2 | 2
  RSV+PIV2 | 1 | 1 | 2
  RSV+PIV3 | 1 | 1 | 2
  RSV+FLUA | 2 | 0 | 2
  RSV+hCOV | 1 | 0 | 1
  HBoV+hCOV | 0 | 1 | 1
  hMPV+hCOV | 1 | 0 | 1
  hCOV+hAV | 1 | 1 | 2
  RSV+HBoV | 1 | 0 | 1
  HRV+FLUA | 0 | 1 | 1
  HRV+HBoV | 1 | 0 | 1
  No virus | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time Taken to Reach the Normal Range for Heart Rate (Per-protocol Analysis)
Description: The time that heart rate takes into the normal range for age between the groups (Per-protocol analysis).
Time Frame: through study completion, an average of 96 hours
Population: The population of the per-protocol.
Measure: Median (Inter-Quartile Range); unit: hour
Groups:
- St-FMOT: Children who received Standard Face Mask Oxygen Therapy
- HFNCOT: Children who received High-Flow Nasal Cannula Oxygen Therapy
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 38 | 38
hour | 12 [2 to 24] | 2 [1 to 4]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Time Taken to Reach the Normal Range for Respiratory Rate (Per-protocol Analysis)
Description: The time that the respiratory rate takes into the normal range for age between the groups (Per-protocol analysis).
Time Frame: through study completion, an average of 96 hours
Population: The population of the per-protocol.
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 38 | 38
hour | 24 [4 to 48] | 4 [2 to 12]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Time Taken to Regress A Lower Clinical Respiratory Score (Per-protocol Analysis)
Description: Unabbreviated scale title: Clinical Respiratory Score (Per-protocol analysis). The time that takes from severe bronchiolitis (9-12 points) to moderate bronchiolitis (5-8 points) or from moderate bronchiolitis (5-8 points) to mild bronchiolitis (0-4 points) between the groups. Higher scores mean a worse outcome. The score ranges from 0-12.
Time Frame: through study completion, an average of 96 hours
Population: The population of the per-protocol.
Measure: Median (Inter-Quartile Range); unit: hour
Groups:
- HFNCT: Children who received High-Flow Nasal Cannula Oxygen Therapy
Arm/Group | St-FMOT | HFNCT
Number analyzed (Participants) | 38 | 38
hour | 4 [2 to 24] | 2 [1 to 4]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCT; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Heart Rate (Intention-to-treat Analysis)
Description: Any differences in the time any recorded changes in heart rate from randomization to the patients' discharge within the groups and between the groups (Intention-to-treat analysis).
Time Frame: Baseline, 1,2,4,12,24,48,72 and 96 hours
Population: Intention to treat analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
beats per minute
  Baseline | 172.90 [167.68 to 178.64] | 171.05 [165.26 to 176.84]
  1 hour | 166.21 [160.99 to 171.43] | 151.28 [145.49 to 157.07]
  2 hours | 164.00 [158.78 to 169.22] | 146.59 [140.80 to 152.38]
  4 hours | 159.65 [154.43 to 164.86] | 138.05 [132.26 to 143.84]
  12 hours | 153.43 [147.88 to 158.98] | 132.47 [126.64 to 138.29]
  24 hours | 142.96 [137.25 to 148.67] | 132.56 [126.71 to 138.40]
  48 hours | 139.21 [133.42 to 145.00] | 128.48 [122.63 to 134.34]
  72 hours | 135.99 [130.09 to 141.90] | 124.96 [118.92 to 130.99]
  96 hours | 133.61 [127.60 to 139.62] | 119.47 [113.15 to 125.80]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p < 0.001, Mixed Models Analysis — The p-Value of the interaction between time and groups was given. In all analyses, p values <0·05 were considered being statistically significant; Mean Difference (Net) = -12.29, 95% CI 2-sided [-23.53 to -1.05], Standard Deviation 5.72 — Treatment difference= High-Flow Nasal Cannula Oxygen Therapy (96-0 h) - Standard Face Mask Oxygen Therapy (96-0 h) (based on least-square means)

5. Secondary Outcome: Heart Rate (Per-protocol Analysis)
Description: Any differences in the time any recorded changes in heart rate from randomization to the patients' discharge within the groups and between the groups (Per-protocol analysis).
Time Frame: Baseline, 1,2,4,12,24,48,72 and 96 hours
Population: Per-protocol analysis
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 38 | 38
beats per minute
  Baseline | 169.03 [164.22 to 173.83] | 170.37 [165.56 to 175.17]
  1 hour | 160.76 [155.96 to 165.57] | 150.37 [145.56 to 155.17]
  2 hours | 157.58 [152.77 to 162.38] | 145.39 [140.59 to 150.20]
  4 hours | 150.66 [145.85 to 155.46] | 136.42 [131.62 to 141.23]
  12 hours | 147.08 [142.27 to 151.88] | 131.32 [126.51 to 136.54]
  24 hours | 138.45 [133.64 to 143.25] | 131.74 [126.93 to 136.54]
  48 hours | 135.97 [131.17 to 140.78] | 127.89 [123.09 to 132.70]
  72 hours | 136.43 [131.54 to 141.31] | 124.57 [119.60 to 129.54]
  96 hours | 133.85 [128.90 to 138.81] | 122.53 [117.30 to 127.76]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; The p-Value of the interaction between time and groups was given. In all analyses, p values <0·05 were considered being statistically significant; Test type: Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -12.66, 95% CI 2-sided [-22.05 to -3.28], Standard Deviation 4.77 — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Respiratory Rate (Intention-to-treat Analysis)
Description: Any differences in the time any recorded changes in respiratory rate from randomization to the patients' discharge within the groups and between the groups (Intention-to-treat analysis).
Time Frame: Baseline, 1,2,4,12,24,48,72 and 96 hours
Population: Intention to treat analysis.
Measure: Median (95% Confidence Interval); unit: Breaths per minute
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
Breaths per minute
  Baseline | 65.08 [62.77 to 67.39] | 66.71 [64.15 to 69.27]
  1 hour | 60.20 [57.89 to 62.51] | 56.84 [54.28 to 59.40]
  2 hours | 57.45 [55.14 to 59.76] | 51.10 [48.54 to 53.66]
  4 hours | 55.54 [53.23 to 57.85] | 46.56 [44.00 to 49.12]
  12 hours | 51.06 [48.63 to 53.48] | 44.15 [41.57 to 46.72]
  24 hours | 46.54 [44.05 to 49.03] | 40.82 [38.24 to 43.40]
  48 hours | 41.89 [39.36 to 44.42] | 39.32 [36.74 to 41.91]
  72 hours | 39.24 [36.65 to 41.82] | 36.70 [34.07 to 39.34]
  96 hours | 37.75 [35.12 to 40.38] | 35.47 [32.79 to 38.22]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p < 0.001, Mixed Models Analysis — The p-Value of the interaction between time and groups was given. In all analysis, p values <0.05 were considered being statistically significant; Mean Difference (Net) = -3.91, 95% CI 2-sided [-8.68 to 0.86], Standard Deviation 2.43 — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Respiratory Rate (Per-protocol Analysis)
Description: Any differences in the time any recorded changes in respiratory rate from randomization to the patients' discharge within the groups and between the groups (Per-protocol analysis).
Time Frame: Baseline, 1,2,4,12,24,48,72 and 96 hours
Population: Per-protocol analysis.
Measure: Median (95% Confidence Interval); unit: breaths per minute
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 38 | 38
breaths per minute
  Baseline | 65.52 [63.15 to 67.89] | 66.68 [64.31 to 69.05]
  1 hour | 59.50 [57.12 to 61.87] | 56.60 [54.23 to 58.97]
  2 hours | 55.34 [52.96 to 57.71] | 50.65 [48.28 to 53.03]
  4 hours | 51.81 [49.44 to 54.18] | 46.00 [43.62 to 48.37]
  12 hours | 48.13 [45.75 to 50.50] | 43.71 [41.33 to 46.08]
  24 hours | 44.23 [41.86 to 46.60] | 40.47 [38.10 to 42.84]
  48 hours | 40.07 [37.70 to 42.45] | 39.05 [36.68 to 41.42]
  72 hours | 37.82 [35.42 to 40.22] | 36.51 [34.09 to 38.92]
  96 hours | 36.63 [34.20 to 39.06] | 35.37 [32.85 to 37.89]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; The p-Value of the interaction between time and groups was given. In all analysis, p values <0.05 were considered being statistically significant; Test type: Other; p = 0.003, Mixed Models Analysis; Mean Difference (Net) = -2.41, 95% CI 2-sided [-6.62 to 1.78], Standard Deviation 2.14 — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Clinical Respiratory Score (Intention-to-treat Analysis)
Description: Unabbreviated scale title: Clinical Respiratory Score (Intention-to-treat analysis) Any differences in the time any recorded changes in the clinical respiratory score from randomization to the patients' discharge within the groups and between the groups.
  This clinical respiratory score includes respiratory rate, retraction, dyspnea/consciousness status, and wheezing.
  The severity of parameters is scored 0 to 3 points, and the patients with a clinical respiratory score of 0-4 points were defined as mild, moderate (5-8 points), and severe (9-12 point) bronchiolitis. Higher scores mean a worse outcome. The score ranges from 0-12.
Time Frame: Baseline, 1,2,4,12,24,48,72 and 96 hours
Population: Intention to treat analysis.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
score on a scale
  Baseline | 9.0 [7.0 to 10.0] | 10.0 [9.0 to 11.0]
  1 hour | 8.0 [6.5 to 10.0] | 7.0 [7.0 to 9.0]
  2 hours | 8.0 [6.0 to 10.0] | 6.0 [5.0 to 8.0]
  4 hours | 7.0 [6.0 to 9.5] | 5.0 [4.0 to 7.0]
  12 hours | 5.0 [4.0 to 7.0] | 5.0 [3.0 to 6.0]
  24 hours | 4.5 [3.0 to 6.0] | 4.0 [2.0 to 5.0]
  48 hours | 3.5 [2.0 to 5.0] | 2.0 [1.0 to 4.0]
  72 hours | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  96 hours | 1.0 [0.0 to 3.0] | 1.0 [0.0 to 2.0]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.002, Brunner-Langer Method — [p-value comment as in outcome 6, analysis 1]; Relative treatment effect difference = -0.07 — Relative Treatment Effect Difference= High-Flow Nasal Cannula Oxygen Therapy (96-0 h) - Standard Face Mask Oxygen Therapy (96-0 h) (based on least-square means)

9. Secondary Outcome: Clinical Respiratory Score (Per-protocol Analysis)
Description: Unabbreviated scale title: Clinical Respiratory Score (Per-protocol analysis). Any differences in the time any recorded changes in the clinical respiratory score from randomization to the patients' discharge within the groups and between the groups. This clinical respiratory score includes respiratory rate, retraction, dyspnea/consciousness status, and wheezing. The severity of parameters is scored 0 to 3 points, and the patients with a clinical respiratory score of 0-4 points were defined as mild, moderate (5-8 points), and severe (9-12 point) bronchiolitis. Higher scores mean a worse outcome. The score ranges from 0-12.
Time Frame: Baseline, 1,2,4,12,24,48,72 and 96 hours
Population: Per-protocol analysis.
Measure: Median (95% Confidence Interval); unit: score on a scale
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 38 | 38
score on a scale
  Baseline | 9.0 [7.0 to 10.2] | 9.5 [8.7 to 11.0]
  1 hour | 8.0 [6.0 to 9.0] | 7.0 [7.0 to 9.0]
  2 hours | 7.0 [5.7 to 8.0] | 6.0 [5.0 to 8.0]
  4 hours | 6.0 [5.0 to 8.0] | 5.0 [4.0 to 6.2]
  12 hours | 5.0 [4.0 to 7.0] | 5.0 [3.0 to 6.0]
  24 hours | 4.5 [2.7 to 6.0] | 4.0 [2.0 to 5.0]
  48 hours | 3.5 [2.0 to 5.0] | 2.0 [1.0 to 4.0]
  72 hours | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  96 hours | 1.0 [0.0 to 3.0] | 1.0 [0.0 to 2.0]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.001, Brunner-Langer Method — [p-value comment as in outcome 6, analysis 1]; Relative treatment effect difference = -0.08 — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Oxygen Requirement (Intention-to-treat Analysis)
Description: The total duration of oxygen therapy (Intention-to-treat analysis).
Time Frame: through study completion, an average of 168 hours
Population: Intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
hour | 29.5 [14.0 to 45.7] | 19.0 [4.0 to 30.0]

11. Secondary Outcome: Oxygen Requirement (Per-protocol Analysis)
Description: The total duration of oxygen therapy (Per-protocol analysis).
Time Frame: through study completion, an average of 168 hours
Population: Per-protocol analysis.
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 38 | 38
hour | 24.0 [12.0 to 38.5] | 18.5 [4.0 to 30.0]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.08, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Length of Hospital Stay (Intention-to-treat Analysis)
Description: The time from randomization to the patient's discharge (Intention-to-treat analysis).
Time Frame: through study completion, an average of 168 hours
Population: Intention to treat analysis.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
day | 5.5 [4.0 to 7.7] | 5.0 [4.0 to 7.0]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.22, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Length of Hospital Stay (Per-protocol Analysis)
Description: The time from randomization to the patient's discharge (Per-protocol analysis).
Time Frame: through study completion, an average of 168 hours
Population: Per-protocol analysis
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 38 | 38
day | 5 [4 to 6] | 5 [4 to 7]
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.99, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Treatment Failure at 4 Hours (Intention-to-treat Analysis)
Description: The number of treatment failures at 4 hours in each study arm (Intention-to-treat analysis).
Time Frame: 4 hours
Population: The population of the intention to treat.
Measure: Count of Participants; unit: Participants
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
Participants | 10 | 1
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.02, Fisher Exact

15. Secondary Outcome: Pediatric Intensive Care Unit Admission (Intention-to-treat Analysis).
Description: The number of participants admitted to the intensive care unit for invasive mechanical ventilation (Intention-to-treat analysis).
Time Frame: through study completion, an average of 168 hours
Population: Intention to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
Participants | 10 | 1
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.02, Fisher Exact

16. Secondary Outcome: Adverse Events of Therapy (Intention-to-treat Analysis)
Description: The number of participants with any adverse events in therapy groups (Intention-to-treat analysis).
Time Frame: through study completion, an average of 168 hours
Population: Intention to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | St-FMOT | HFNCOT
Number analyzed (Participants) | 48 | 39
Participants | 1 | 5
Statistical Analysis 1: Comparison: St-FMOT vs HFNCOT; Test type: Other; p = 0.08, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 6 weeks.
Groups:
- Active Comparator: High-Flow Nasal Cannula Oxygen Therapy: Children in the high-flow group received heated and humidified high-flow oxygen at a rate of 2 L*kg/min (maximum 25 L/min), using an age-appropriate Optiflow Junior cannula and Airvo 2 high-flow system (Fisher and Paykel Healthcare). The initial fraction of inspired oxygen (FiO2) was set at 40%. The starting flow rate continued for a minimum of 4 hours. According to the patients' clinical response, the flow rate was decreased by 0.5 L*kg/min per hour. The FiO2 was adjusted to obtain the oxygen saturation levels between 92-98%. When the flow rate was at 0.5 L*kg/min, and the FiO2 was equal to the ambient oxygen concentration, High-Flow nasal cannula oxygen therapy was stopped.
- Active Comparator: Standard Face Mask Oxygen Therapy: Children in the standard-therapy group received supplemental oxygen via a simple face mask, a range of 6-10 L/min, to maintain the oxygen saturation level between 92-98%. Those who sustained the oxygen saturation >92% in the ambient oxygen concentration were weaned off Standard Face Mask Oxygen Therapy.
Arm/Group | Active Comparator: High-Flow Nasal Cannula Oxygen Therapy | Active Comparator: Standard Face Mask Oxygen Therapy
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/48
Other Adverse Events (participants affected / at risk) | 5/39 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: High-Flow Nasal Cannula Oxygen Therapy (N=39) | Active Comparator: Standard Face Mask Oxygen Therapy (N=48)
Transient bradicardia (Cardiac disorders) | 3 | 1
Epistaxis (General disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was performed in a single center and had a limited sample size. We did not blind the allocation of oxygen therapies to introduce the risk of performance bias.

We did not reach the number of participants calculated with the power analysis because of the financial support problem. Therefore, we used effect size for each of the primary outcomes.

Patients were not allocated to receive therapy in a ratio of 1:1. Hence, a numerical difference occurred between the two groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT04245202/Prot_SAP_000.pdf